CLINICAL TRIAL: NCT05770921
Title: An Exploratory Study of Pulsed Field Ablation Device and Force Sensing Pulsed Field Ablation Catheter Guided by Columbus 3D EP Navigation System in the Ablation Treatment of Paroxysmal Supraventricular Tachycardia（PSVT）
Brief Title: Pulsed Field Ablation for Paroxysmal Supraventricular Tachycardia（PSVT）
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Principal Investigator, Caijie Shen, Director, Ningbo No. 1 Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 775035
Record Dates: First submitted 2023-01-30; First posted 2023-03-16 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Paroxysmal Supraventricular Tachycardia
Keywords: PSVT; PFA; AVNRT; AVRT
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Intervention Model Description: prospective, single-center, single-group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Non-randomized (Experimental): All subjects will be ablated using the Pulsed Field Ablation Device and Force Sensing Pulsed Field Ablation Catheter in the management of their Paroxysmal Supraventricular Tachycardia
  Interventions: Device: Pulsed Field Ablation Device and Force Sensing Pulsed Field Ablation Catheter

INTERVENTIONS:
Device: Pulsed Field Ablation Device and Force Sensing Pulsed Field Ablation Catheter — All subjects will be ablated using the Pulsed Field Ablation Device and Force Sensing Pulsed Field Ablation Catheter in the management of their Paroxysmal Supraventricular Tachycardia

SUMMARY:
The purpose of this study was to explore the safety and efficacy of a Pulsed Field Ablation Device and Force Sensing Pulsed Field Ablation Catheter in the treatment of Paroxysmal Supraventricular Tachycardia.

DETAILED DESCRIPTION:
The Primary Endpoint for efficacy is the number of subjects where ablation of each PSVT resulted in confirmation of electrical isolation of the PSVT 15 minutes following the last index PFA application with the investigational device

ELIGIBILITY:
Inclusion Criteria:

1. Patients with symptomatic paroxysmal supraventricular tachycardia including:Atrioventricular nodal re-entrant tachycardia, Atrioventricular arrhythmias;
2. Willingness to undergo an evaluation to validate the requirements of the protocol.
3. Voluntary signed informed consent and willingness to undergo the tests and procedures required by the protocol.

Exclusion Criteria:

1. Patients with structural heart disease
2. History of any cardiac surgery
3. Failure of prior ablation of PSVT
4. Presence of any implantation, such as artificial valves, permanent pacemakers, etc
5. Patients with active systemic infections
6. Any condition contraindicating septal puncture or retrograde transaortic approach for procedures
7. Any condition contraindicating heparin or aspirin
8. Patients with advanced malignant tumor
9. Any woman known to be pregnant or breastfeeding
10. Unwilling or unable to comply fully with study procedures and follow-up
11. Unable to provide own informed consent
12. Coexistence with other arrhythmias

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-07-13 (Actual)

PRIMARY OUTCOMES:
Immediate ablation success rate | 15 minutes post ablation
  The Primary Endpoint for efficacy is the number of subjects where ablation of each PSVT resulted in confirmation of electrical isolation of the PSVT 15 minutes following by catheter mapping and ECG to determine immediate ablation success rate
Rate of Treatment Success at 6-Month Post-Procedure | Refers to the postoperative phase after 6 months postoperatively
  Refers to the postoperative phase after 6 months follow-up after process,by ECG, Holter, or Heart rate monitoring method based on equivalent confirmed that there are no PSVT events account for the number of participants into the group of the proportion of the total number.

SECONDARY OUTCOMES:
Rate of Treatment Success at 1-Month Post-Procedure | Refers to the postoperative phase after 1 months postoperatively
  Refers to the postoperative phase after 1 months follow-up after process,by ECG, Holter, or Heart rate monitoring method based on equivalent confirmed that there are no PSVT events account for the number of participants into the group of the proportion of the total number.
Rate of Treatment Success at 2-Month Post-Procedure | Refers to the postoperative phase after 2 months postoperatively
  Refers to the postoperative phase after 2 months follow-up after process,by ECG, Holter, or Heart rate monitoring method based on equivalent confirmed that there are no PSVT events account for the number of participants into the group of the proportion of the total number.
Evaluation of Force Sensing Pulsed Field Ablation Catheter | 1 Day of surgery
  Evaluation of catheter operation performance;Catheter ablation parameters
Evaluation of Pulse Ablation equipment | immediately post ablation
  System software operability; System operation stability; Hardware connection validity

OTHER OUTCOMES:
Security Endpoints | Within 6 months after sign the informed consent form
  Incidence of adverse events and serious adverse events associated with the study device

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shen C, Du X, Dai J, Feng M, Yu Y, Liu J, Fu G, Wang B, Jiang Y, Jin H, Chu H. Outcomes of Focal Pulsed Field Ablation for Paroxysmal Supraventricular Tachycardia. Can J Cardiol. 2024 Jul;40(7):1294-1303. doi: 10.1016/j.cjca.2023.12.037. Epub 2024 Jan 17. PMID 38242530